CLINICAL TRIAL: NCT03593980
Title: Gastric Emptying Following an Oral Carbohydrate Load in Women Admitted for Elective Cesarean Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study could not be run for logistical reasons
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-06
Record Dates: First submitted 2018-06-27; First posted 2018-07-20 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Pregnancy; Respiratory Aspiration of Gastric Contents
Keywords: Gastric Ultrasound
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 400ml cranberry juice (Experimental): Patients will be given 400ml of cranberry juice to drink 3 hours prior to cesarean delivery.
  Interventions: Dietary Supplement: Cranberry juice

INTERVENTIONS:
Dietary Supplement: Cranberry juice — 400ml cranberry juice

SUMMARY:
Because of the risk of pulmonary aspiration, patients are asked to comply with the fasting guidelines when they are scheduled for an elective cesarean section. This fasting can result in increased insulin resistance, and that this can delay patient recovery from surgery. Giving a patient a carbohydrate-rich beverage before surgery has been shown to reduce the post-operative insulin resistance and reduce the length of stay in the hospital.

In order to safely provide pregnant women with a carbohydrate-rich drink when admitted to the hospital in preparation for an elective cesarean delivery, the investigators must ensure that their stomach has emptied by the time they go to the operating room.

The objective is to investigate whether women admitted to the hospital, having complied with the fasting guidelines, will have an empty stomach 2 hours after being offered 400 ml of a beverage containing 50g of carbohydrate. This can easily be done with the use of an ultrasound exam of the stomach.

The hypothesis is that patients will have an empty stomach 2 hours after drinking 400 ml of a carbohydrate-rich beverage.

DETAILED DESCRIPTION:
Fasting, even if for brief periods, results in a marked reduction in insulin sensitivity. This insulin resistance developed after surgery has been implicated in the increase of the length of stay at the hospital. Randomized studies involving either preoperative glucose infusion or ingestion of a carbohydrate-rich beverage have shown that postoperative insulin resistance may be reduced by about 50% when preoperative fasting is avoided.

One of the recommended methods to avoid the insulin resistance in the perioperative period is the provision of isotonic, carbohydrate-containing clear fluids up to 2 hours preoperatively, so that patients begin their surgery in a fed rather than fasted state. This has been called "carbohydrate loading". An amount of 50 g of carbohydrates is sufficient to produce an insulin response similar to that of a mixed solid meal.

Beverages containing different combinations of carbohydrate or protein have been used in different patient populations and support the safety of their use in the perioperative period. Although there is substantial evidence that gastric emptying is similar in non-laboring term pregnant women and non-pregnant it is unknown whether the maternal anxiety preceding the procedure and the addition of a 50 g carbohydrate containing beverage may cause delayed gastric emptying and increase the risk of aspiration in the obstetric population.

Bedside ultrasound assessment of the gastric content has shown good intra- and inter-rater reliability. Our group has previously demonstrated that in 103 women scheduled for elective cesarean, 95% of fasting subjects presented with an antral cross-sectional area ≤10.3 cm2.

In order to implement and to standardize a beverage containing 50 g of complex carbohydrate offered to women when admitted to the hospital in preparation for their elective cesarean delivery, the investigators must ensure that women have an empty stomach by the time they arrive to the operating room.

ELIGIBILITY:
Inclusion Criteria:

* non-laboring pregnant women ≥36 weeks gestational age, scheduled for cesarean delivery
* ≥18 years of age
* ASA physical status II to III
* weight 50 to 120 kg
* height ≥150 cm
* ability to understand the rationale of the study assessments.

Exclusion Criteria:

* Diabetes Mellitus
* patients who have not complied with fasting guidelines (8 hours of solid food or thick fluids, and no clear fluid 3 hours before the scheduled arrival time on Labor and Delivery for the study)
* abnormal anatomy of the upper gastrointestinal tract, and previous surgical procedures on the esophagus, stomach, or upper abdomen
* gastric ultrasound that is not compatible with empty stomach (gastric antrum grade 0 or 1 and CSA < 10.3 cm2 in the right lateral decubitus).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Antral cross sectional area 2 hours | 2 hours
  The antral cross sectional area will be measured using ultrasound at 2 hours after consumption of a 400ml beverage

SECONDARY OUTCOMES:
Qualitative assessment of the antrum | 2 hours
  The antrum will be viewed and graded (0-2, where 0=empty, 1=fluid and 2=solid/mixed meal content) at 5 minutes, 1 hour and 2 hours after consumption of a 400ml beverage
Antral cross sectional area at 5 min | 5 min
  The antral cross sectional area will be measured using ultrasound at 5 minutes after consumption of a 400ml beverage
Antral cross sectional area at 1 hour | 1hour
  The antral cross sectional area will be measured using ultrasound at 1 hour after consumption of a 400ml beverage
Patient satisfaction | 2 hours
  Patient satisfaction will be assessed in the immediate postoperative period, on a Likert scale from 1-5 (1=strongly disagree and 5=strongly agree)
Intraoperative hypotension | 1 hour
  Blood pressure during surgery measuring less than 80% of the patient's baseline
Presence of intraoperative pain | 1 hour
  Pain will be self reported by the patient and treated by the physicians taking care of them.
  Patients may be asked to rate their pain on a 0-10 scale (where 0 is no pain and 10 is the most terrible pain). Pain during surgery that requires opioid supplementation (at the discretion of the attending physician) will be considered.
Presence of intraoperative nausea: questionnaire (yes/no) | 1 hour
  Patients will be asked to report any nausea during surgery. This will be recorded as 0=no presence of nausea, or 1=presence of nausea.
Presence of intraoperative vomiting: (yes/no) | 1 hour
  Vomiting at any time during the surgery will be recorded (where 0=no vomiting, and 1=presence of vomiting).

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada